CLINICAL TRIAL: NCT03116568
Title: A Prospective Study of Pregnant Women With and Without IBD in Order to Better Understand the Patterns of Bacterial Transmission From the Mother to the Baby (Bacterial Transmission In Utero and IBD Risk)
Brief Title: Bacterial Transmission In Utero and IBD Risk
Status: Active, not recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Siew Chien NG, Professor, Chinese University of Hong Kong
Other Study IDs: The Meconium Study
Record Dates: First submitted 2017-04-12; First posted 2017-04-17 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: IBD; Pregnancy Related; Microbiota
Keywords: IBD; Meconium; Pregnancy; Microbiota; Newborn

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool, meconium, placenta, saliva and cord blood.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IBD Case: 1. Pregnant women with IBD
  2. Newborns of pregnant women with IBD
  3. Family member of pregnant women with IBD
  4. Siblings of newborns
- Control: 1. Pregnant women without IBD
  2. Newborns of pregnant women without IBD
  3. Family member of pregnant women without IBD
  4. Siblings of newborns

SUMMARY:
Inflammatory bowel diseases (IBD), Crohn's disease (CD) and ulcerative colitis (UC), are caused by the loss of mucosal tolerance towards the commensal microbiota resulting in inflammatory responses.

Identifying intestinal bacteria in mother and newborn of both IBD and Control groups allow us to understand the change of bacterial composition human microbiome in the gut during pregnancy and childhood development.

DETAILED DESCRIPTION:
Inflammatory bowel diseases (IBD), Crohn's disease (CD) and ulcerative colitis (UC), are caused by the loss of mucosal tolerance towards the commensal microbiota resulting in inflammatory responses.

Human microbiome studies have demonstrated dynamic changes in bacterial composition in the gut during pregnancy and childhood development. Moreover, the presence of pathogenic species, or absence of beneficial species, in early childhood has been suggested to play a key role in the initiation of preterm birth, development of asthma or eczema, allergy, autism or other immunological deficiency. The goal of this study is to better understand the link between maternal and newborn microbiome. Specifically, we will investigate the microbial composition of the stool of newborn babies born to mothers with certain health issues as compared to healthy mothers. This information may help identify the factors that can help better understand the risk transmitted through the microbiome.

By collecting the samples including stools, saliva and understanding the health history of pregnant women with or without Inflammatory bowel disease (IBD), we can compare the data of two groups pregnant women in order to find out the differences of microbiome in their guts. Another aim of our study is finding out the possibility of vertical bacteria transmission from mother to baby.

Furthermore, our main focus is the meconium of newborn baby, we would like to know that the differences of microbiome in the gut between the newborns from two groups. Therefore, we will collect the umbilical cord blood, placenta, amniotic membrane, newborn cheek swab, and meconium. To investigate the disease transmission rate from mothers.

ELIGIBILITY:
1. Pregnant Women with IBD (Case) Inclusion Criteria 1. Be pregnant or planning pregnancy 2. To have confirmed IBD 3. To plan giving birth in Hong Kong Exclusion Criteria 1. Pregnancy complications, such as intrauterine fetal demise/stillbirth, preeclampsia, hyperemesis gravidarum, active infection, including chorioamnionitis or sepsis 2. Fetus chromosomal or structural abnormalities 3. Known history of HIV 4. History of Colectomy or ileo-anal pouch
2. Pregnant Women without IBD (Control) Inclusion Criteria 1. To be pregnant or planning pregnancy 2. Subjects without IBD 3. To plan giving birth in Hong Kong Exclusion Criteria 1. Pregnancy complications, such as intrauterine fetal demise/stillbirth, preeclampsia, hyperemesis gravidarum, active infection, including chorioamnionitis or sepsis 2. Fetus chromosomal or structural abnormalities 3. Known history of HIV 4. History of colectomy or ileo-anal pouch 5. Autoimmune diseases 6. Blood in stools 7. History of perianal fistula or abscesses
3. Family Members Inclusion Criteria 1. Residing in the same household with the pregnant woman from both case and control groups e.g. child, spouse, parents of the pregnant woman 2. The subject or, when applicable, the subject's legally acceptable representative (or parent or legal guardians) signs and dates a written, informed consent form prior to the initiation of study.
4. New Born Baby Inclusion Criteria 1. Be a new born baby of enrolled pregnant women from both case and control groups 2. The subject's parents or legally guardians sign and date a written, informed consent form prior to the initiation of study.

Max Age: 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects include (1) pregnant women with IBD (case), (2) pregnant women without IBD (control), (3) family members of pregnant women from both groups and (4) new born baby of both groups
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2017-04-24 (Actual); Primary Completion 2025-04-14 (Estimated); Study Completion 2027-09-27 (Estimated)

PRIMARY OUTCOMES:
Relation of microbiota in the gut between mother and new-borns | 5 years after the mother give birth
  Identify different type of intestial bacteria between both IBD and Control groups

CONTACTS AND LOCATIONS:
Overall Officials: Siew Chien Ng, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong